CLINICAL TRIAL: NCT01199289
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Determine the Safety and Efficacy of AMG 827 in Subjects With Inadequately Controlled Asthma
Brief Title: A Study to Evaluate the Dosing of AMG 827 for Subjects With Inadequately Controlled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20090203
Record Dates: First submitted 2010-08-05; First posted 2010-09-10 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Amgen; chronic inflammatory disease; wheezing
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive the matching placebo administered as subcutaneous (SC) injections at Day 1 and weeks 1, 2, 4, 6, 8, and 10.
  Interventions: Drug: Placebo
- AMG 827 140 mg (Experimental): Participants will receive AMG 140 mg administered as SC injections at Day 1 and weeks 1, 2, 4, 6, 8, and 10.
  Interventions: Drug: AMG 827
- AMG 827 210 mg (Experimental): Participants will receive AMG 210 mg administered as SC injections at Day 1 and weeks 1, 2, 4, 6, 8, and 10.
  Interventions: Drug: AMG 827
- AMG 827 280 mg (Experimental): Participants will receive AMG 280 mg administered as SC injections at Day 1 and weeks 1, 2, 4, 6, 8, and 10.
  Interventions: Drug: AMG 827

INTERVENTIONS:
Drug: AMG 827 — SC injection.
  Arms: AMG 827 140 mg; AMG 827 210 mg; AMG 827 280 mg
Drug: Placebo — SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if AMG 827 is effective compared to placebo as measured by change in Asthma Control Questionnaire (ACQ) composite scores.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 65 years of age
* Percent of predicted FEV1 ≥ 50% and ≤ 80%
* At least 12% reversibility over pre-bronchodilator FEV1
* Inhaled corticosteroid (ICS) ≥ 200 and ≤ 1000 µg/day fluticasone powder or equivalent
* Ongoing asthma symptoms with ACQ composite score ≥ 1.5 points

Exclusion Criteria:

* Respiratory infection within 4 weeks of screening visit or 1 week of baseline visit
* History of chronic obstructive pulmonary disease or other chronic pulmonary condition other than asthma
* Any uncontrolled or clinically significant systemic disease (eg, uncontrolled diabetes, liver disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2010-10-04 (Actual); Primary Completion 2011-12-21 (Actual); Study Completion 2011-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (49):
- United States (22):
  - Research Site, Encinitas, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Stockton, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Stockbridge, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Bozeman, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Skillman, New Jersey
  - Research Site, Rockville Centre, New York
  - Research Site, High Point, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Lake Oswego, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Madison, Wisconsin
- Austria (3):
  - Research Site, Feldbach
  - Research Site, Hallein
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Turku
- Hungary (5):
  - Research Site, Edelény
  - Research Site, Mátraháza
  - Research Site, Tatabánya
  - Research Site, Törökbálint
  - Research Site, Zalaegerszeg - Pozva
- Research Site, Rotterdam, Netherlands
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Chodzież
  - Research Site, Gdansk
  - Research Site, Wroclaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Korea (3):
  - Research Site, Bucheon-si
  - Research Site, Seoul
  - Research Site, Suwon

REFERENCES:
- [Background] Busse WW, Holgate S, Kerwin E, Chon Y, Feng J, Lin J, Lin SL. Randomized, double-blind, placebo-controlled study of brodalumab, a human anti-IL-17 receptor monoclonal antibody, in moderate to severe asthma. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1294-302. doi: 10.1164/rccm.201212-2318OC. PMID 24200404
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 61 centers in Austria, Belgium, Canada, Finland, Hungary, Netherlands, Poland, Russia, South Korea, and the United States; 47 of these sites enrolled participants from 04 October 2010 to 21 December 2011. 315 participants were enrolled, but 10 participants from 1 site were excluded from all analyses due to major issues of Good Clinical Practice (GCP) compliance and are not included in the participant flow.
Pre-assignment Details: A washout period for specific asthma medications was conducted after informed consent and prior to run-in period. After completing screening and meeting all eligibility criteria, all eligible participants underwent run-in visits for 4 weeks prior to randomization.
Groups:
- Placebo: Participants received the matching placebo administered as a subcutaneous (SC) injection at Day 1 and weeks 1, 2, 4, 6, 8, and 10.
- AMG 827 140 mg: Participants received AMG 827 140 mg administered as a SC injection at Day 1 and weeks 1, 2, 4, 6, 8, and 10.
- AMG 827 210 mg: Participants received AMG 872 210 mg administered as a SC injection at Day 1 and weeks 1, 2, 4, 6, 8, and 10.
- AMG 827 280 mg: Participants received AMG 827 280 mg administered as a SC injection at Day 1 and weeks 1, 2, 4, 6, 8, and 10.
Period: Overall Study
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Started | 77 | 75 | 76 | 77
Participants Who Received Study Treatment | 76 | 74 | 76 | 76
Completed | 68 | 68 | 71 | 65
Not Completed | 9 | 7 | 5 | 12
Not completed — Ineligibility determined | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Noncompliance | 1 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 3 | 1 | 4
Not completed — Full consent withdrawn | 2 | 2 | 2 | 3
Not completed — Administrative decision | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol-specified criteria | 3 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least 1 dose of study treatment and were not excluded from analysis due to GCP violations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg | Total
Number analyzed (Participants) | 76 | 74 | 76 | 76 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (11.2) | 43.6 (11.6) | 46.0 (11.2) | 46.5 (11.5) | 45.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 42 | 38 | 46 | 179
  Male | 23 | 32 | 38 | 30 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 6 | 3 | 20
  Not Hispanic or Latino | 73 | 66 | 70 | 73 | 282
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 55 | 63 | 67 | 254
  Black or African American | 5 | 16 | 6 | 4 | 31
  Asian | 2 | 3 | 2 | 3 | 10
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Multiple | 0 | 0 | 2 | 2 | 4
  Other | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Composite Scores to Week 12
Description: The ACQ is an instrument used in clinical research and practice to evaluate asthma control/impairment.
  It is a validated composite score that assesses disease control by evaluating 7 questions: night time awakenings, asthma symptoms upon awakening, activity limitation, shortness of breath, wheeze frequency, short-acting bronchodilator use, and forced expiratory volume in 1 second (FEV1).
  The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/limitation) scale. The total score is obtained by adding the value from each question and dividing by the number of questions. Higher scores indicates worsening of condition and a negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: All randomized participants who received at least 1 dose of study treatment who were not excluded due to GCP violations, and had non-missing baseline and post-baseline data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 76 | 73 | 75 | 74
Score on a scale | -0.427 (0.784) | -0.521 (0.796) | -0.512 (0.728) | -0.556 (0.810)
Statistical Analysis 1: Comparison: Placebo vs AMG 827 140 mg; Test type: Superiority; p = 0.5838, ANCOVA; LS Mean Difference = -0.068, 95% CI 2-sided [-0.311 to 0.175]
Statistical Analysis 2: Comparison: Placebo vs AMG 827 210 mg; Test type: Superiority; p = 0.5391, ANCOVA; LS Mean Difference = -0.075, 95% CI 2-sided [-0.316 to 0.166]
Statistical Analysis 3: Comparison: Placebo vs AMG 827 280 mg; Test type: Superiority; p = 0.3583, ANCOVA; LS Mean Difference = -0.113, 95% CI 2-sided [-0.355 to 0.129]

2. Secondary Outcome: Change From Baseline in Pre- and Post-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. FEV1 was performed both pre and post-administration of bronchodilator treatment at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 76 | 73 | 75 | 74
Liters (L)
  Pre-Bronchodilator | 0.075 (0.323) | 0.035 (0.307) | 0.066 (0.367) | 0.058 (0.348)
  Post-Bronchodilator: number analyzed (Participants) | 70 | 65 | 70 | 67
  Post-Bronchodilator | -0.052 (0.275) | -0.019 (0.259) | 0.016 (0.227) | -0.032 (0.285)
Statistical Analysis 1: Comparison: Placebo vs AMG 827 140 mg; Pre-Bronchodilator; Test type: Superiority; p = 0.4076, ANCOVA; LS Mean Difference = -0.047, 95% CI 2-sided [-0.157 to 0.064]
Statistical Analysis 2: Comparison: Placebo vs AMG 827 210 mg; Pre-Bronchodilator; Test type: Superiority; p = 0.6915, ANCOVA; LS Mean Difference = -0.022, 95% CI 2-sided [-0.130 to 0.086]
Statistical Analysis 3: Comparison: Placebo vs AMG 827 280 mg; Pre-Bronchodilator; Test type: Superiority; p = 0.7271, ANCOVA; LS Mean Difference = -0.019, 95% CI 2-sided [-0.126 to 0.088]
Statistical Analysis 4: Comparison: Placebo vs AMG 827 140 mg; Post-Bronchodilator; Test type: Superiority; p = 0.9210, ANCOVA; LS Mean Difference = 0.005, 95% CI 2-sided [-0.086 to 0.095]
Statistical Analysis 5: Comparison: Placebo vs AMG 827 210 mg; Post-Bronchodilator; Test type: Superiority; p = 0.1139, ANCOVA; LS Mean Difference = 0.070, 95% CI 2-sided [-0.017 to 0.157]
Statistical Analysis 6: Comparison: Placebo vs AMG 827 280 mg; Post-Bronchodilator; Test type: Superiority; p = 0.6426, ANCOVA; LS Mean Difference = 0.021, 95% CI 2-sided [-0.066 to 0.107]

3. Secondary Outcome: Change From Baseline in AM and PM Peak Expiratory Flow Rate (PEFR) to Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litres/minute
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 76 | 74 | 76 | 75
Litres/minute
  AM | 4.26 (39.220) | -14.09 (46.708) | -4.53 (46.468) | -1.95 (44.624)
  PM | -0.22 (37.807) | -11.56 (40.277) | -9.16 (45.080) | -7.96 (37.984)
Statistical Analysis 1: Comparison: Placebo vs AMG 827 140 mg; AM; Test type: Superiority; p = 0.0262, ANCOVA; LS Mean Difference = -16.847, 95% CI 2-sided [-31.686 to -2.009]
Statistical Analysis 2: Comparison: Placebo vs AMG 827 210 mg; AM; Test type: Superiority; p = 0.3627, ANCOVA; LS Mean Difference = -6.723, 95% CI 2-sided [-21.239 to 7.793]
Statistical Analysis 3: Comparison: Placebo vs AMG 827 280 mg; AM; Test type: Superiority; p = 0.4507, ANCOVA; LS Mean Difference = -5.488, 95% CI 2-sided [-19.791 to 8.814]
Statistical Analysis 4: Comparison: Placebo vs AMG 827 140 mg; PM; Test type: Superiority; p = 0.1228, ANCOVA; LS Mean Difference = -10.426, 95% CI 2-sided [-23.686 to 2.834]
Statistical Analysis 5: Comparison: Placebo vs AMG 827 210 mg; PM; Test type: Superiority; p = 0.3092, ANCOVA; LS Mean Difference = -6.738, 95% CI 2-sided [-19.758 to 6.281]
Statistical Analysis 6: Comparison: Placebo vs AMG 827 280 mg; PM; Test type: Superiority; p = 0.2167, ANCOVA; LS Mean Difference = -8.043, 95% CI 2-sided [-20.831 to 4.744]

4. Secondary Outcome: Change From Baseline in the Frequency of Rescue Short Acting β-Agonist (SABA) Use to Week 12
Description: Participants recorded SABA use for 1 week prior to randomization (baseline) and the average number of days recorded was subtracted from average days of SABA use across 12 week intervention period.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 76 | 74 | 76 | 75
Days | -0.630 (2.842) | -0.187 (2.971) | -0.727 (2.941) | -0.798 (4.293)
Statistical Analysis 1: Comparison: Placebo vs AMG 827 140 mg; Test type: Superiority; p = 0.5157, ANCOVA; LS Mean Difference = 0.331, 95% CI 2-sided [-0.670 to 1.332]
Statistical Analysis 2: Comparison: Placebo vs AMG 827 210 mg; Test type: Superiority; p = 0.6434, ANCOVA; LS Mean Difference = -0.234, 95% CI 2-sided [-1.229 to 0.760]
Statistical Analysis 3: Comparison: Placebo vs AMG 827 280 mg; Test type: Superiority; p = 0.6954, ANCOVA; LS Mean Difference = -0.199, 95% CI 2-sided [-1.196 to 0.799]

5. Secondary Outcome: Change From Baseline in Daily Asthma Symptom Score to Week 12
Description: Participants recorded their daily asthma symptoms in their electronic diaries (Ediary). It included 7 questions: frequency of night time awakening, time awake at night, wheezing, shortness of breath, cough, chest tightness and activity limitation.
  Daily asthma symptoms score is the sum of 7 individual scores (with the total score ranging from 0-21).
  Higher scores indicates worsening of condition and a negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 76 | 74 | 76 | 75
Score on a scale | -1.531 (3.674) | -1.816 (3.250) | -1.629 (2.620) | -1.607 (3.238)
Statistical Analysis 1: Comparison: Placebo vs AMG 827 140 mg; Test type: Superiority; p = 0.5577, ANCOVA; LS Mean Difference = -0.283, 95% CI 2-sided [-1.231 to 0.665]
Statistical Analysis 2: Comparison: Placebo vs AMG 827 210 mg; Test type: Superiority; p = 0.9366, ANCOVA; LS Mean Difference = 0.038, 95% CI 2-sided [-0.904 to 0.980]
Statistical Analysis 3: Comparison: Placebo vs AMG 827 280 mg; Test type: Superiority; p = 0.7745, ANCOVA; LS Mean Difference = 0.138, 95% CI 2-sided [-0.808 to 1.084]

6. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Score at Week 12
Description: The AQLQ is the most commonly used asthma specific instrument and includes evaluations of both symptom and quality of life measures. The 32-item instrument measures 4 domains affected by asthma including activity limitations, emotional function, exposure to environmental stimuli, and symptoms (Mitchell EA et al, 1997, Juniper et al, 1994, Christie MJ et al, 1993, Juniper et al, 1993).
  Participants were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (7=no impairment, 1=severe impairment). The overall score = mean of the responses to the 32 questions.
  Higher scores indicate "better quality of life" and a positive change from baseline indicates improved symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 66 | 65 | 69 | 63
Score on a scale | 0.626 (0.901) | 0.596 (0.979) | 0.537 (0.710) | 0.587 (0.866)
Statistical Analysis 1: Comparison: Placebo vs AMG 827 140 mg; Test type: Superiority; p = 0.8524, ANCOVA; LS Mean Difference = 0.026, 95% CI 2-sided [-0.251 to 0.303]
Statistical Analysis 2: Comparison: Placebo vs AMG 827 210 mg; Test type: Superiority; p = 0.8139, ANCOVA; LS Mean Difference = -0.033, 95% CI 2-sided [-0.305 to 0.240]
Statistical Analysis 3: Comparison: Placebo vs AMG 827 280 mg; Test type: Superiority; p = 0.9881, ANCOVA; LS Mean Difference = -0.002, 95% CI 2-sided [-0.281 to 0.276]

7. Secondary Outcome: Proportion of Asthma Symptom-free Days
Description: Asthma symptom-free days were defined as a participant having a score of zero in their daily asthma symptom score. Asthma symptom-free days without SABA use were defined as a participant having a score of zero in their daily asthma symptom score and no SABA use.
  The proportion of asthma symptom-free days was calculated as the number of asthma symptom-free days over the number of days in the double-blind treatment period (12 weeks).
Time Frame: Up to Week 12
Population: All randomized participants who received at least 1 dose of study treatment who were not excluded due to GCP violations
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 76 | 74 | 76 | 76
Ratio
  With use of SABA | 0.230 (0.299) | 0.167 (0.263) | 0.198 (0.293) | 0.166 (0.267)
  Without use of SABA | 0.201 (0.294) | 0.123 (0.241) | 0.181 (0.286) | 0.146 (0.256)
Statistical Analysis 1: Comparison: Placebo vs AMG 827 140 mg; Test type: Superiority — With use of SABA; p = 0.1213, ANCOVA; LS Mean Difference = -0.062, 95% CI 2-sided [-0.141 to 0.017]
Statistical Analysis 2: Comparison: Placebo vs AMG 827 210 mg; Test type: Superiority — With use of SABA; p = 0.6643, ANCOVA; LS Mean Difference = -0.017, 95% CI 2-sided [-0.095 to 0.061]
Statistical Analysis 3: Comparison: Placebo vs AMG 827 280 mg; Test type: Superiority; p = 0.2879, ANCOVA; With use of SABA; LS Mean Difference = -0.042, 95% CI 2-sided [-0.121 to 0.036]
Statistical Analysis 4: Comparison: Placebo vs AMG 827 140 mg; Test type: Superiority — Without use of SABA; p = 0.0546, ANCOVA; LS Mean Difference = -0.074, 95% CI 2-sided [-0.150 to 0.001]
Statistical Analysis 5: Comparison: Placebo vs AMG 827 210 mg; Without use of SABA; Test type: Superiority; p = 0.9078, ANCOVA; LS Mean Difference = -0.004, 95% CI 2-sided [-0.080 to 0.071]
Statistical Analysis 6: Comparison: Placebo vs AMG 827 280 mg; Without use of SABA; Test type: Superiority; p = 0.3616, ANCOVA; LS Mean Difference = -0.035, 95% CI 2-sided [-0.111 to 0.040]

8. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of AMG 827 at Week 8 to 10
Time Frame: Week 8 (days 60 and 64), and pre-dose on Week 10
Population: The pharmacokinetic (PK) analyses set: all participants who received at least one dose of AMG 827 and who had at least 1 PK concentration measurement.
Measure: Median (Full Range); unit: Days
Arm/Group | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 33 | 35 | 29
Days | 3.1 [0.0 to 8.0] | 3.1 [0.0 to 9.1] | 3.9 [1.9 to 13.0]

9. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 827 at Week 8 to 10
Time Frame: Week 8 (days 60 and 64), and pre-dose on Week 10
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 33 | 35 | 29
µg/mL | 8.11 (6.91) | 16.6 (12.4) | 29.4 (17.5)

10. Secondary Outcome: Area Under the Concentration-time Curve During the Dosing Interval (AUCtau) of AMG 827 at Week 8 to 10
Time Frame: Week 8 (days 60 and 64), and pre-dose on Week 10
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
Number analyzed (Participants) | 33 | 35 | 29
µg*day/mL | 68.3 (74.3) | 171 (150) | 313 (196)

ADVERSE EVENTS:
Time Frame: Day 1 to Week 16
Description: All-cause mortality is reported for all participants randomized in the study that were not excluded from analysis due to GCP violations. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug that were not excluded from analysis due to GCP violations.
Arm/Group | Placebo | AMG 827 140 mg | AMG 827 210 mg | AMG 827 280 mg
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/75 | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/76 | 3/74 | 1/76 | 2/76
Other Adverse Events (participants affected / at risk) | 24/76 | 28/74 | 28/76 | 28/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | AMG 827 140 mg (N=74) | AMG 827 210 mg (N=76) | AMG 827 280 mg (N=76)
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Degeneration of uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | AMG 827 140 mg (N=74) | AMG 827 210 mg (N=76) | AMG 827 280 mg (N=76)
Injection site erythema (General disorders) | 2 | 5 | 7 | 7
Nasopharyngitis (Infections and infestations) | 5 | 5 | 3 | 3
Oral candidiasis (Infections and infestations) | 0 | 1 | 4 | 3
Sinusitis (Infections and infestations) | 4 | 2 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 8 | 4 | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 18 | 15 | 14
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 4

LIMITATIONS AND CAVEATS:
10 participants from 1 site were excluded from all analysis due to major GCP violations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.